CLINICAL TRIAL: NCT03138187
Title: Effect of Physical Exercise Intensity on Spontaneous Physical Activity Energy Expenditure and Energy Intake in Overweight Adults: a Study Protocol for a Randomized Controlled Trial.
Brief Title: Physical Exercise and Energy Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Rosely Sichieri, Full professor, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: exercise and obesity
Record Dates: First submitted 2017-04-30; First posted 2017-05-03 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Physical Activity
Keywords: spontaneous physical activity; caloric intake
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants and physical trainer blinding will not be feasible due to the characteristics of prescribed exercise sessions. However, the evaluators will be blinded to the following endpoints: weight, body composition, appetite, energy intake and laboratorial biomarkers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (No Intervention): without physical exercise sessions
- Moderate exercise group (Experimental): The training phase of the moderate exercise group (MEG) will consist of 4 sets of 10 minutes walking/running at moderate intensity, with 5 minutes walking at low intensity for recovery between sets
  Interventions: Behavioral: Moderate exercise
- Vigorous exercise group (Experimental): The training phase of the vigorous exercise group (VEG) will consist of 4 sets of 10 minutes running at vigorous intensity, with 5 minutes walking at low intensity for recovery between sets
  Interventions: Behavioral: Vigorous exercise

INTERVENTIONS:
Behavioral: Moderate exercise — The training phase of the moderate exercise group (MEG) will consist of 4 sets of 10 minutes walking/running at moderate intensity, with 5 minutes walking at low intensity for recovery between sets
  Arms: Moderate exercise group
Behavioral: Vigorous exercise — The training phase of the vigorous exercise group (VEG) will consist of 4 sets of 10 minutes running at vigorous intensity, with 5 minutes walking at low intensity for recovery between sets
  Arms: Vigorous exercise group

SUMMARY:
This study is a randomized controlled trial, designed to evaluate the effect of structured physical exercise sessions on the spontaneous physical activity energy expenditure and caloric intake in overweight adults. The design employs a parallel three-group experimental arms: (1) a moderate exercise group (MEG); (2) a vigorous exercise group (VEG); and a control group (CG) without physical exercise sessions.

ELIGIBILITY:
Inclusion Criteria:

1. male
2. overweight

Exclusion Criteria:

1. diabetes mellitus
2. cardiovascular diseases
3. musculoskeletal injuries

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — only male
Enrollment: 72 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
spontaneous physical activity energy expenditure | 15 days
  Physical activity energy expenditure will be assessed by a triaxial accelerometers (ActiGraph GT3x-BT, Pensacola, FL, USA). The device will be positioned at the anterior axillary line of the non-dominant hip, for 15 consecutive days

SECONDARY OUTCOMES:
appetite sensations | 15 days
  Subjective hunger and satiety sensations will be measured through the visual analog scale (VAS) proposed by Flint et al. (2000).
energy intake | 15 days
  Food and beverages consumption will be assessed by 24-h food recalls (REC24h). Nutritionists will conduct a face-to-face interview in four different moments during the intervention period: at the 2nd and 5th days (Tuesday and Friday) in the first week; and at the 11th and 15th days (Thursday and Monday) in the second week, including weekdays and weekend.
laboratorial biomarkers | 15 days
  To investigate the physiological mechanisms involved in energy expenditure and food consumption regulation, blood and salivary samples will be collected to biochemical and hormonal analyses at the 1st (baseline) and the 15th days of the intervention period, in the morning, after at least 10 hours of fasting.

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Academy, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paravidino VB, Mediano MFF, Crochemore-Silva I, da Cruz VL, Antunes MML, Beaulieu K, Gibbons C, Finlayson G, Blundell JE, Sichieri R. The compensatory effect of exercise on physical activity and energy intake in young men with overweight: The EFECT randomised controlled trial. Physiol Behav. 2021 Feb 1;229:113249. doi: 10.1016/j.physbeh.2020.113249. Epub 2020 Nov 20. PMID 33221391
- [Derived] Paravidino VB, Mediano MFF, Silva ICM, Wendt A, Del Vecchio FB, Neves FA, Terra BS, Gomes EAC, Moura AS, Sichieri R. Effect of physical exercise on spontaneous physical activity energy expenditure and energy intake in overweight adults (the EFECT study): a study protocol for a randomized controlled trial. Trials. 2018 Mar 7;19(1):167. doi: 10.1186/s13063-018-2445-6. PMID 29514690